CLINICAL TRIAL: NCT03492021
Title: The Role of Beef in Optimal Protein and Feeding Strategies to Accelerate Muscle Mass and Functional Recovery From Anterior Cruciate Ligament (ACL) Repair
Brief Title: Protein in Feeding Strategies to Accelerate Muscle Recovery From ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Orthopedic Associates of Hartford (Unknown); United States Army Research Institute of Environmental Medicine (U.S. Federal Agency); University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Nancy Rodriguez, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HHC-E-HHC-2016-0126; KFS63669550 (Other Grant/Funding Number: National Cattlemen's Beef Association)
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Rehabilitative Nutrition for Muscle Recovery From ACL Reconstruction
Keywords: rehabilitative nutrition; protein; beef; ACL reconstruction; protein synthesis; proteolysis; muscle mass; muscle strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adequate Protein_Carbohydrate Post Therapy (Experimental): Diet Intervention - Adequate Protein (1.0 g/kg/d) - Carbohydrate Post Therapy [AP-CPT]
  Interventions: Other: Diet Intervention_AP-CPT
- Optimal Protein_Protein Post Therapy (Experimental): Diet Intervention - Optimal Protein (2.0 g/kg/d) - Protein Post Therapy [OP-PPT]
  Interventions: Other: Diet Intervention_PP-PPT

INTERVENTIONS:
Other: Diet Intervention_AP-CPT — Adequate Protein_Carbohydrate Post Therapy (AP-CPT) where protein intake will be 1 g/kg/d for the duration of the study .
  Arms: Adequate Protein_Carbohydrate Post Therapy
Other: Diet Intervention_PP-PPT — Optimal Protein_Protein Post Therapy (OP-PPT) with protein intake set at 2.0 g/kg/day for the duration of the study
  Arms: Optimal Protein_Protein Post Therapy

SUMMARY:
Musculoskeletal injury, particularly injuries requiring surgical repair, induce significant muscle atrophy, resulting in diminished physical function. The protein turnover-associated (diminished protein synthesis, elevated protein breakdown, negative net muscle protein balance) etiology of injury and surgical-induced atrophy are, in part, similar to those observed with muscle wasting induced by hyper-catabolic and inflammatory conditions and prolonged periods of skeletal muscle disuse (e.g., cachexia and joint immobilization). Combining dietary strategies to optimize the anabolic properties of beef as a high quality protein source that provides essential amino acids prior to surgery and throughout post-surgery rehabilitation may attenuate muscle atrophy and accelerate the restoration of muscle function. This project will examine the efficacy of habitual consumption of a beef-based higher protein meal pattern and post-physical rehabilitation beef protein supplementation throughout post-surgical rehabilitation intervention on skeletal muscle function in response to anterior cruciate ligament (ACL) repair in healthy, physically active adults.

Stable isotope methodologies, proteomic analysis of muscle protein synthesis, and molecular assessments of skeletal muscle atrophy and remodeling will be assessed to evaluate the effects of increased protein intake, including consumption of a high quality beef-based protein supplement following patient physical therapy sessions on:

1. Skeletal muscle protein fractional synthetic rates during and in recovery from surgery;
2. Inflammatory, proteolytic, and anabolic intramuscular signaling during surgery and their association with skeletal muscle protein synthesis and muscle function;
3. Muscle size and functional recovery;
4. Duration to return to routine exercise, sport, or physical activity.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age
* identified as appropriate for study recruitment by their respective orthopedic surgeon
* undergoing their first anterior cruciate ligament (ACL) repair
* undergo ACL reconstruction under general anesthesia
* body mass indexes (BMIs) within normal to overweight ranges

Exclusion Criteria:

* reporting metabolic or cardiovascular abnormalities, food allergies, gastrointestinal disorders (i.e. lactose intolerance)
* use of nutritional/herbal/sports supplements including anabolic steroids, and tobacco products will be excluded from the study
* BMIs above 29.9

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle protein fractional synthetic rates | Following 16 weeks of physical rehabilitation post surgery for subjects in both diet intervention groups.
  Using stable isotope techniques skeletal muscle protein fractional synthetic rates will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R Rodriguez, PhD, Principal Investigator — University of Connecticut-Storrs
Locations (1):
- Orthopedic Associates of Hartford, Hartford, Connecticut, United States